CLINICAL TRIAL: NCT06376721
Title: A Phase Ib/II Clinical Trial of Linperlisib Combined With Camrelizumab and Pegaspargase in Advanced or Relapsed/Refractory NK/T-cell Lymphoma
Brief Title: Linperlisib Combined With Camrelizumab and Pegaspargase in Advanced or Relapsed/Refractory NK/T-cell Lymphoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Principal Investigator, LIANG WANG, Director of the department of hematology, Beijing Tongren Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TREC2024-KY016
Record Dates: First submitted 2024-04-15; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Natural Killer/T-Cell Lymphoma, Nasal and Nasal-Type; T-lymphoblastic Lymphoma
Keywords: r/r ENKTL; Linperlisib; PD-1 blockade; Pegaspargase
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — camrelizumab; Injections; pegaspargase; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Treatment with linperlisib in combination with camrelizumab and pegaspargase for advanced or relapsed/refractory ENKTCL patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment arm (Experimental): Linperlisib:
  Phase Ib：oral, 80 mg/d, QD; Phase II： oral, RP2D, QD.
  Camrelizumab for Injection:
  Phase Ib & Phase II：intravenous drip, 200 mg/d, Q3W, administered on day 1 of each cycle (3 weeks in each cycle)
  Pegaspargase:
  Phase Ib & Phase II：intramuscular injection，2500 IU/m2, Q3W, administered on day 1 of each cycle (3 weeks in each cycle)
  Interventions: Drug: Linperlisib; Drug: Camrelizumab; Drug: Pegaspargase; Drug: Dexamethasone

INTERVENTIONS:
Drug: Linperlisib — Linperlisib: Phase Ib, oral, 80 mg/d, QD; Phase II, oral, RP2D, QD.
  Other Names: YY-20394
Drug: Camrelizumab — Camrelizumab for Injection: 200 mg/d, intravenous drip for 30 min (not less than 20 min and not more than 60 min), administered on day 1 of each cycle, observed for 2 hours after infusion. Every 3 weeks is a dosing cycle. Cycle 2 and subsequent cycles of dosing may be administered up to 5 days before or after the day of the scheduled dosing; more than 3 days after the date of the scheduled dosing will be considered a delayed dosing.
  Other Names: Camrelizumab for Injection
Drug: Pegaspargase — Pegaspargase: 2500 IU/m2, intramuscular injection, divided into three places, administered on the first day of each cycle, observed 2 hours after injection for the occurrence of anaphylactic reaction, if there is no anaphylactic reaction before giving other test drugs. Every 3 weeks as a dosing cycle.
  Camrelizumab for Injection should not be applied on the same day as Dexamethasonee.
  Other Names: Pegaspargase injection
Drug: Dexamethasone — Dexamethasone, 20 mg/d, days 1-4. Camrelizumab for Injection should not be applied on the same day as Dexamethasonee.
  Other Names: Dexamethasone oral

SUMMARY:
The patients diagnosed with relapsed/refractory or advanced NK/T-cell Lymphoma (r/r NKTCL) were selected as the research objects. To explore effective and safe treatment for advanced or r/r NKTCL, the combination of PI3K-δ inhibitor Linperlisib with PD-1 blockade Camrelizumab and anti-metabolic agent Pegaspargase was applied for the treatment.

DETAILED DESCRIPTION:
This is a prospective, single-arm, single-center Ib/II clinical trial that included an initial safety run-in phase with safety monitoring before the main enrollment (expansion phase).The aim of phase Ib is to evaluate the recommended phase 2 dose and dose-limiting toxicity (DLT), and the aim of phase II study is to evaluate, for the first time, the safety and efficacy of the treatment of Linperlisib combined with PD-1 blockade Camrelizumab and Pegaspargase in patients diagnosed with advanced or r/r ENKTL, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Histopathology and immunohistochemistry confirmed diagnosis of ENKTL according to WHO 2016 criteria.
* refractory or relapsed after initial remission, or Ann-Arbor stage III-IV de novo patients
* PET/CT or CT/MRI with at least one objectively evaluable lesion.
* Expected to survive more than 3 months.
* General status ECOG score 0-2 points.
* The laboratory test within 1 week before enrollment meets the following conditions:

Blood routine: WBC≥3×10e9/L, PLT≥75×10e9/L, ANC≥1.5×10e9/L. sCR≤1.5 mg/dL,GFR≥50 ml/min. Liver function: ALT & AST≤3 times the upper limit of normal, TBIL ≤2 times the upper limit of normal.

Serum fibrinogen level≥1.0 g/L.

•Sign the informed consent form

Exclusion Criteria:

* Patients with CNS involvement, or with other neoplasm;
* Patients has received PI3K inhibitor treatment before enrollment
* Poor performance status, ECOG≥2;
* Patients in lactation or pregnancy；
* Patients (male or female) have the possibility of childbirth but are unwilling or have not taken effective contraceptive measures；
* Patients allergic to any of the study drugs；
* Patients with active infection；
* Patients with a history of immunodeficiency, including HIV positive or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation;
* Patients with a history of interstitial pneumonia, non infectious pneumonia, or highly suspected interstitial pneumonia;
* Patients with a history of neurological or psychiatric disorders, including epilepsy or dementia, in the past
* According to the researcher's judgment, there are accompanying diseases that seriously endanger patient safety or affect patient completion of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2024-04-14 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
The best objective response rate（ORR） over 6 treatment cycles | Within 6 treatment cycles (each cycle is 21 days)
  Overall response rate means sum of complete response rate and partial response rate

SECONDARY OUTCOMES:
Objective Response Rate（ORR） | At the end of 2nd, 4th, 6th treatment cycles,respectively (each cycle is 21 days)
  Objective response rate means sum of complete response rate and partial response rate
Complete Response （CR） | At the end of 2nd, 4th, 6th treatment cycles,respectively (each cycle is 21 days)
  CR was defined as complete remission evaluated using PET-CT scan or BM test
Progression Free Survival (PFS) | From date of enrollment until the date of progression or date of death from any cause, whichever came first, assesed up to 2 years.
  Progression free survival was defined as the period from the start of treatment to the date of confirmed disease progression or death from any cause.
Overall Survival (OS) | From date of enrollment until the date of documented death from any cause or follow up, whichever came first, assesed up to 2 years.
  Overall survival is defined as the time from the date of treatment to the date of death.
Disease Control Rate（DCR） | Up to 2 years after enrollment.
  Disease control rate discribes the percentage of patients with advanced cancer whose therapeutic intervention has led to a complete response, partial response, or stable disease

OTHER OUTCOMES:
Drug safety | up to 2 years after enrollment
  According to NCI CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Liang Wang, M.D., Principal Investigator — Beijing Tongren Hospital
Locations (1):
- Liang Wang, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No